CLINICAL TRIAL: NCT06389981
Title: Co-Design and Pilot Testing of Peer-led Community Outreach to Improve Equity, Veteran-Centeredness and Uptake of Lung Cancer Screening
Acronym: VPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Renda Wiener, Principal Investigator, VA Boston Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1692052
Record Dates: First submitted 2024-04-01; First posted 2024-04-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer led intervention (Experimental): The peer-led program will be pilot tested enrolling 40 self-identified lung cancer screening eligible Black Veterans.
  Interventions: Other: Veterans peer connect Program

INTERVENTIONS:
Other: Veterans peer connect Program — To assess outcomes of the Peer-led program, the study team will collect information from Veteran pilot test participants via surveys and data abstraction on healthcare utilization (Lung cancer screening completion, tobacco treatment) from the Veterans Affairs Corporate Data Warehouse. Survey data will be collected at 3 timepoints: baseline, post-Peer-led orientation, and 3-months post-enrollment. Healthcare utilization data will be abstracted from the corporate data warehouse to reflect the 3-month post-enrollment timepoint. Finally, interviews will be conducted with a subset of participants.

SUMMARY:
Co-design will be implemented to develop an innovative, Veteran-centered intervention (Vet Peer Connects program) that meets the needs of Black Veterans.

Next, a feasibility pilot test of the Vet Peer Connects program will be conducted. The Peer will lead up to 4 group lung cancer screening orientations in community partner sites to reach around 40 lung cancer screening eligible Black Veterans. The Peer will provide one-to-one tailored support to up to 15 Veterans (coaching, goal-setting, navigation to access Veterans Affairs lung cancer screening). Then, the study team will evaluate program delivery through ethnographic observation and field notes, Peer activity logs, and weekly check-ins between the study team and Peer. Investigators will interview Veteran participants, community partners, and lung cancer screening clinical staff to explore feasibility and acceptability of the Vet Peer Connects program and solicit suggestions for improvement. Preliminary data on the outcomes of the Vet Peer Connects program will be collected by study team through administering surveys to assess change in Social Cognitive Theory constructs, and extracting lung cancer screening uptake and tobacco treatment 3 months post enrollment from VA's Corporate Data Warehouse. This work will inform a subsequent multi-site stepped-wedge trial to assess effectiveness, implementation, and cost of the Vet Peer Connects program in VA lung cancer screening sites and neighboring branches of the National Association for Black Veterans

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black Veterans
* Meet United States Preventive Services Task Force guidelines for lung cancer ( still smoking cigarettes or quit within past 15 years, greater than or equal to 20 pack-years total)
* Have not yet undergone lung cancer screening

Exclusion Criteria:

* Non-Black Veterans

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Lung Cancer Screening Uptake | 3 months
  Assessing electronic health record data to determine if screening has occurred

SECONDARY OUTCOMES:
Tobacco cessation Treatment | 3 months
  Assessing electronic health record data to determine if tobacco treatment has been utilized
Stigma Related to Smoking | 7 months
  Assess via qualitative interviews
Perceived support from peer | 7 months
  Assess via qualitative interviews
Lung Cancer Screening Knowledge | 7 months
  Knowledge of risks and benefits of lung cancer screening Scale 0-18, higher score means a better outcome
Lung Cancer Screening Fatalism | 7 months
  Adapted Illness Perception Questionnaire. Scale 10-50, higher score means better outcome
Trust in VA | 7 months
  Adapted Modified trust scale for Veterans Affairs health system New Scale 4-20, higher score means a better outcome
Lung Cancer Self-efficacy | 7 months
  Lung cancer screening health belief self-efficacy scale Scale 9-36, higher score means a better outcome
General Cancer Self-efficacy | 7 months
  New General Self-efficacy scale Scale 8-40, higher score means a better outcome
Intention to engage in shared decision making | 7 months
  Preparation for Decision Making, scale 10-40, lower score means better outcome
Motivation to quit smoking | 7 months
  Readiness to change smoking behavior, contemplation ladder, scale 1-10, higher score means a better outcome
Intention to undergo lung cancer screening | 7 months
  Low Literacy Decisional Conflict Scale Scale 0-9, higher score means a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication. Prior to distribution, a local privacy officer will certify that all datasets contains no protected health information. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by office of research and development. Those requesting data will be asked to sign a Letter of Agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year of publication
Access Criteria: Those requesting data will be asked to sign a Letter of Agreement.